CLINICAL TRIAL: NCT00471939
Title: A Phase II, Multi-Centre, Controlled Study of the Safety and Efficacy of Wound Healing Gel I-020502 (KUR-212) in Patients Undergoing Autologous Meshed Skin Grafting.
Brief Title: Safety and Efficacy of I-020502 in Meshed Skin Autografting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Collaborators: Baxter BioScience (Industry)
Responsible Party: Virginia Jamieson, Kuros Biosurgery AG
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS I-020502/01
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Burns
Keywords: Burn, Meshed skin graft, PDGF; deep partial thickness or full thickness burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: I-020502 — 1 mcg/mL TG-PDGF.AB

SUMMARY:
This is a phase II, multi-centre, controlled study comparing the safety and tolerability on wound healing following an application of I-020502 in a concentration of 1μg/mL TG-PDGF.AB versus staples applied in the same patient to burn areas requiring autologous meshed skin grafting.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by the patient or his/her legal representative.
2. Male or female, aged ≥ 18 years.
3. Female with childbearing potential with a negative pregnancy test within 3 day prior to surgery (screening).
4. Patients with burn wound(s) between ≥ 5 % and ≤ 50 % TBSA.
5. Patients with a contiguous deep partial thickness/full thickness wound(s) of two comparable sites either contiguous or separate in the same location (e.g. leg) each sized between 1% and 2% TBSA but not more than 400 cm2.
6. Patients who are willing to comply with treatment applications and instructions by the protocol.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding.
2. Patients with known or suspected allergies to any of the components of the wound healing gel I-020502 (e.g. hypersensitivity to bovine proteins).
3. Digits, head, genitalia, palms of hands, soles of feet, and face are excluded as test sites.
4. Electrical and/or chemical burns.
5. Patients that are judged to have significant pulmonary compromise.
6. Transcutaneous tissue oxygenation < 90%.
7. Clinically significant infections at wound sites.
8. Clinically significant systemic infections.
9. Suspicion or presence of active systemic or local cancer or tumor of any kind.
10. Patients with known immunodeficiency disorders, either congenital or acquired.
11. Patients with vascular or skin disorders that directly affect the designated wound site.
12. Patients with Diabetes mellitus.
13. Patients with chronic malnourishment.
14. Chronic treatment with immunosuppressive drugs or systemic corticosteroids within the last 2 months prior to surgery.
15. Any other acute or chronic concurrent medical conditions that in the Investigator's opinion are a contraindication to skin mesh grafting and study participation.
16. Participation in another investigational study within 30 days prior to surgery, for investigational devices, or within the last three months for investigational drugs related to wound healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events up to 28 days post surgery | 28 days

SECONDARY OUTCOMES:
Incidence of AE/SAE, Changes in vital signs, Hematology/clinical chemistry, PDGF.AB/TG-PDGF.AB and antibodies, hypergranulation, Percentage and proportion of re-epithelialization/engraftment, Scar assessment, Time and resources for test site treatments | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lehnhardt, Dr., Principal Investigator — Universitätsklinik für Plastische Chirurgie und Schwerbrandverletzte
Locations (1):
- Universitätsklinik für Plastische Chirurgie und Schwerbrandverletzte, Bochum, Germany